CLINICAL TRIAL: NCT07326969
Title: MOVEMENT ANALYSIS IN PATIENTS UNDERGOING VERTEBRECTOMIES FOR THE TREATMENT OF SPINE ONCOLOGY: A PILOT STUDY
Brief Title: MOVEMENT ANALYSIS IN PATIENTS UNDERGOING VERTEBRECTOMIES FOR SPINE ONCOLOGY: A PILOT STUDY
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: GAV
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Spine Tumor; Vertebral Metastasis; Vertebral Column Mass
Keywords: vertebrectomy; gait analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- vertebrectomy: patients with vertebral tumors undergoing vertebrectomy
  Interventions: Other: vertebrectomy

INTERVENTIONS:
Other: vertebrectomy — en bloc resection of oncological vertebra

SUMMARY:
Analyze the geometric and kinematic parameters of the spine in patients undergoing vertebrectomy through gait analysis, both during the execution of motor tasks such as walking, standing, and basic trunk movements, with the aim of improving the assessment and, therefore, possibly, the treatment and the final clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Presence of spinal cancer with surgical indication for vertebrectomy
* Approval and signature of informed consent for the study
* Ability to undergo movement analysis before the surgery and the 6-month follow-up

Exclusion Criteria:

* Under 18 years of age
* Presence of degenerative, traumatic, or infectious pathologies or spinal deformities
* Absence of a signed informed consent form
* Inability to undergo movement analysis before the surgery or the 6-month follow-up

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with vertebral tumors undergoing vertebrectomy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-12-21 (Actual)

PRIMARY OUTCOMES:
Gait Analysis | 6 months after vertebrectomy
  Measure and correlate geometric and kinematic parameters of the trunk and spine through instrumental motion analysis, before and after vertebrectomy surgery in patients with oncological spinal diseases.

SECONDARY OUTCOMES:
questionnaire | 6 months after vertebrectomy
  Evaluate patient-reported functional outcomes through self-administered questionnaires: Oswestry Disability Index and Fall Efficacy Scale-International
spino-pelvic parameters | 6 months after vertebrectomy
  Measure the geometric spino-pelvic parameters (static) and compare them with the kinematic parameters (dynamic)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided